CLINICAL TRIAL: NCT02621307
Title: The Effect of Salba (Salvia Hispanica L) Versus Flax on Postprandial Blood Glucose Response and Subjective Appetite in Healthy Individuals
Brief Title: Effect of Salba & Flax on Postprandial Glycemia and Subjective Satiety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Vladimir Vuksan, Research Scientist & Professor, Unity Health Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GLUSEED
Record Dates: First submitted 2015-11-27; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Hyperglycemia, Postprandial
Keywords: postprandial glycemia; subjective appetite; Salba; Flax
MeSH Terms: conditions — Hyperglycemia | interventions — Linseed Oil; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Salba (Experimental): 50g glucose 25g ground Salba (Salba Corporation Ltd, Buenos Aires, Argentina) 200ml water
  Interventions: Dietary Supplement: Salba
- Flax (Experimental): 50g glucose 31g ground Flax (Bob's Red Mill Natural Raw Whole Flaxseed) 200ml water
  Interventions: Dietary Supplement: Flax
- Control (Placebo Comparator): 50g glucose 200ml water
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Salba
  Other Names: Salvia hispanica L
  Arms: Salba
Dietary Supplement: Flax
  Arms: Flax
Dietary Supplement: Control
  Other Names: Glucose
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether drinks containing Salvia hispanica L (Salba) or Flax lower postprandial blood glucose levels and improve appetite in healthy individuals.

DETAILED DESCRIPTION:
Dietary fibre has been implicated in improving many risk factors associated with Type 2 Diabetes and Cardiovascular Disease (CVD). However, on average, Norther Americans consume less than half of the recommended amount set by health agencies. It has been proposed that the health benefits of dietary fibre may be attritbuted to rheological characteristics such as viscosity. Salvia hispanica L (Salba) and Flax are nutritionally similar. The primary objective of this research trial is to study the effects of Salba and Flax on postprandial glycemia and appetite in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 35 kg/m^2

Exclusion Criteria:

* known history of liver or kidney disease, diabetes, hypertension, stroke, or myocardial infarctions, thyroid disease, gastrointestinal disease, or AIDS
* subjects using medications or Natural Health Products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in Postprandial Blood Glucose | 2 Hours
  At each visit, postprandial blood glucose will be measured via capillary blood samples, at 15, 30, 45, 60, 90, and 120 minutes after intake of test meals

SECONDARY OUTCOMES:
Change in Subjective Satiety | 2 Hours
  At each visit, subjective satiety (how hungry/full you feel) will be measured via questionnaires, at 15, 30, 45, 60, 90, and 120 minutes after intake of test meals

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada